CLINICAL TRIAL: NCT04988503
Title: Bare Platinum Coils Versus Second-generation Hydrocoils for the Endovascular Treatment of Ruptured Intracranial Aneurysms: a Randomized Controlled Study
Brief Title: Bare Platinum Coils Versus Second-generation Hydrocoils
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to HEC supply issues at participating centers and low enrollment rate among eligible patients
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pusan National University Yangsan Hospital (Other); Chungnam National University Sejong Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2012/652-002
Record Dates: First submitted 2021-07-23; First posted 2021-08-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Aneurysm, Ruptured; Intracranial Aneurysm
Keywords: aneurysms; embolization; rupture
MeSH Terms: conditions — Aneurysm, Ruptured; Intracranial Aneurysm; Aneurysm; Rupture

STUDY DESIGN:
Intervention Model Description: bare platinum coils group versus second-generation hydrogel coil group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Second-generation hydrogel coil group (Experimental): Treatment using second-generation hydrogel coils (had to constitute > 50% of the total coil length) for ruptured cerebral aneurysms
  Interventions: Device: Coil embolization
- Bare platinum coil group (Active Comparator): Treatment using bare metal coil only for ruptured cerebral aneurysms
  Interventions: Device: Coil embolization

INTERVENTIONS:
Device: Coil embolization — coil embolization for ruptured intracranial aneurysm with bare platinum coils or second-generation hydrogel coils

SUMMARY:
Comparison of clinical and radiological outcomes between bare platinum coil group and second-generation hydrogel coils for treatment of ruptured intracranial aneurysms.

DETAILED DESCRIPTION:
The investigators aimed to analyze whether the use of second-generation hydrogel coils for the treatment of ruptured intracranial aneurysms improves clinical and angiographic outcomes compared with the use of bare platinum coils.

ELIGIBILITY:
Inclusion Criteria:

* 19 year old or older
* untreated ruptured intracranial aneurysms with an anatomy such that endovascular treatment with either bare platinum or second-generation hydrogel coils was considered feasible.
* person who agreed to study

Exclusion Criteria:

* contrast allgery (+)
* combined other intracranial lesions (tumor, moyamoya disease, cerebral vascular diseases)
* ineligible for coil embolization

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
any recurrence rate after treatment | during 12 months after coil embolization
  any recurrence rate at 12 months after coil embolization

SECONDARY OUTCOMES:
rate of retreatment during 12 months follow-up period | rate of retreatment during 12 months follow-up period
  rate of retreatment during 12 months follow-up period
packing density (%) after coil embolization | packing density (%) after coil embolization
  packing density (%) after coil embolization
Procedural complication | during coil embolization
  Procedural complication
delayed cerebral ischemia during 12-month follow-up period | delayed cerebral ischemia during 12-month follow-up period
  delayed cerebral ischemia during 12-month follow-up period
good clinical outcome (mRS score ≤ 2) at 12-month follow-up period | good clinical outcome (mRS score ≤ 2) at 12-month follow-up period
  good clinical outcome (mRS score ≤ 2) at 12-month follow-up period
rate of ventriculoperitoneal shunt during 12-month follow-up period | rate of ventriculoperitoneal shunt during 12-month follow-up period
  rate of ventriculoperitoneal shunt during 12-month follow-up period
coil's ease of manipulation | during coil embolization
  coil's ease of manipulation

CONTACTS AND LOCATIONS:
Overall Officials: O-Ki Kwon, Principal Investigator — Seoul National University Bundang Hospital
Locations (3):
- South Korea (3):
  - Chungnam National University Sejong Hospital, Sejong, Chungcheongnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Seoul National University Bundang Hospital, Seongnam-si

IPD SHARING:
Plan to Share IPD: No